CLINICAL TRIAL: NCT00821379
Title: Complications of PCOS Pregnancy: Evaluating Risk
Brief Title: CoPPer Study - Complications of Polycystic Ovary Syndrome (PCOS) Pregnancy: Evaluating Risk
Acronym: CoPPer
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: The Queen Elizabeth Hospital (Other); Erasmus Medical Center (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: UMC Utrecht, Department of Obstetrics and Gynaecology
Other Study IDs: CoPPer study - 07/331; NL 20244.041.07 (ABR)
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2009-01

CONDITIONS: Pregnancy Complications; Delivery Complications; Neonatal Complications
Keywords: PCOS; Polycystic Ovary Syndrome; Pregnancy Complications; Gestational Diabetes; Pre eclampsia; Prediction Model; Pre conceptional
MeSH Terms: conditions — Pregnancy Complications; Polycystic Ovary Syndrome; Diabetes, Gestational; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum and lithium heparine, urine and placenta tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The CoPPer study is a follow-up study of women diagnosed with Polycystic Ovary Syndrome (PCOS). Women will be included pre-conceptional and followed-up until after delivery. The investigators will design a multivariate prediction model of pregnancy outcome in women with PCOS with the intention to define intervention strategies for the future.

DETAILED DESCRIPTION:
Background of the study:

PCOS is a heterogeneous condition in which metabolic disturbances such as insulin resistance are common. Pregnancies in women with PCOS are reported to have an increased chance of being complicated by gestational diabetes, pregnancy induced hypertension and pre-eclampsia. Subsequently their offspring are reported to have a lower birth weight and higher risk of admission to a neonatal intensive care unit. However, the cause of increased complication rate is not yet identified.

There is evidence that intra-uterine conditions as well as pre- and periconception factors influence not only neonatal outcome, but also long-term health of the child. Therefore early detection and treatment of pregnancy complications is important for both mother and child.

In order to identify high risk PCOS pregnancies, the specific effects of PCOS on pregnancy in comparison to the background effects need further investigation.

Preconceptional risk assessment of PCOS women is needed to improve antenatal health care and pregnancy outcome of PCOS pregnancies in the future.

Objective of the study:

To design a multivariate prediction model of pregnancy outcome in women with PCOS with the intention to define intervention strategies for the future.

Study design:

Prospective multi-centre follow-up cohort study.

Method:

Women with PCOS will be screened and included in the study pre-conceptionally. Endocrinological values, glucose tolerance and ultrasound scan etc will be recorded. During pregnancy, blood samples will be stored regularly and glucose measurement will be done. Post-partum the pregnancy outcome will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS
* 18 to 40 years old, who wish to conceive.

Exclusion Criteria:

* Women with anovulation that is not caused by PCOS
* Women with a language barrier
* Women under 18 or over 40 years of age will be excluded from participation.

Other exclusion criteria are:

* Unresolved medical conditions
* Established type 1 diabetes.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with PCOS and a wish to conceive who attend to the University Hospital in Utrecht.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart CJ Fauser, MD PhD, Study Director — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Christ JP, Gunning MN, Meun C, Eijkemans MJC, van Rijn BB, Bonsel GJ, Laven JSE, Fauser BCJM. Pre-Conception Characteristics Predict Obstetrical and Neonatal Outcomes in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2019 Mar 1;104(3):809-818. doi: 10.1210/jc.2018-01787. PMID 30590587
- [Derived] de Wilde MA, Lamain-de Ruiter M, Veltman-Verhulst SM, Kwee A, Laven JS, Lambalk CB, Eijkemans MJC, Franx A, Fauser BCJM, Koster MPH. Increased rates of complications in singleton pregnancies of women previously diagnosed with polycystic ovary syndrome predominantly in the hyperandrogenic phenotype. Fertil Steril. 2017 Aug;108(2):333-340. doi: 10.1016/j.fertnstert.2017.06.015. PMID 28778282
- [Derived] Daan NM, Koster MP, Steegers-Theunissen RP, Eijkemans MJ, Fauser BC. Endocrine and cardiometabolic cord blood characteristics of offspring born to mothers with and without polycystic ovary syndrome. Fertil Steril. 2017 Jan;107(1):261-268.e3. doi: 10.1016/j.fertnstert.2016.09.042. Epub 2016 Oct 27. PMID 28228318
- [Derived] Koster MP, de Wilde MA, Veltman-Verhulst SM, Houben ML, Nikkels PG, van Rijn BB, Fauser BC. Placental characteristics in women with polycystic ovary syndrome. Hum Reprod. 2015 Dec;30(12):2829-37. doi: 10.1093/humrep/dev265. Epub 2015 Oct 25. PMID 26498178
- [Derived] de Wilde MA, Goverde AJ, Veltman-Verhulst SM, Eijkemans MJ, Franx A, Fauser BC, Koster MP. Insulin action in women with polycystic ovary syndrome and its relation to gestational diabetes. Hum Reprod. 2015 Jun;30(6):1447-53. doi: 10.1093/humrep/dev072. Epub 2015 Apr 2. PMID 25840428
- [Derived] de Wilde MA, Veltman-Verhulst SM, Goverde AJ, Lambalk CB, Laven JS, Franx A, Koster MP, Eijkemans MJ, Fauser BC. Preconception predictors of gestational diabetes: a multicentre prospective cohort study on the predominant complication of pregnancy in polycystic ovary syndrome. Hum Reprod. 2014 Jun;29(6):1327-36. doi: 10.1093/humrep/deu077. Epub 2014 Apr 28. PMID 24777850
- [Derived] Veltman-Verhulst SM, Goverde AJ, van Haeften TW, Fauser BC. Fasting glucose measurement as a potential first step screening for glucose metabolism abnormalities in women with anovulatory polycystic ovary syndrome. Hum Reprod. 2013 Aug;28(8):2228-34. doi: 10.1093/humrep/det226. Epub 2013 Jun 5. PMID 23739218
- [Derived] Veltman-Verhulst SM, Fauser BC, Eijkemans MJ. High singleton live birth rate confirmed after ovulation induction in women with anovulatory polycystic ovary syndrome: validation of a prediction model for clinical practice. Fertil Steril. 2012 Sep;98(3):761-768.e1. doi: 10.1016/j.fertnstert.2012.04.027. Epub 2012 May 24. PMID 22633255
- [Derived] Veltman-Verhulst SM, van Haeften TW, Eijkemans MJ, de Valk HW, Fauser BC, Goverde AJ. Sex hormone-binding globulin concentrations before conception as a predictor for gestational diabetes in women with polycystic ovary syndrome. Hum Reprod. 2010 Dec;25(12):3123-8. doi: 10.1093/humrep/deq272. Epub 2010 Oct 13. PMID 20943702